CLINICAL TRIAL: NCT04427644
Title: Is Body Mass Index and Obesity Surgery Mortality Risk Score Important in Perioperative Complications of Laparoscopic Sleeve Gastrectomy Before Discharge? A Retrospective Cohort Study
Brief Title: Body Mass Index and Obesity Surgery Mortality Risk Score in Perioperative Complications of Laparoscopic Sleeve Gastrectomy
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Mehmet Buğra Bozan, Professor, Assistant, Kahramanmaras Sutcu Imam University
Other Study IDs: 13281952-929
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Perioperative Complication; Laparascopic Sleeve Gastrectomy; BMD; Obesity, Morbid; Obesity Surgery Mortality Score; Clavien Dindo Surgical Complication Scale
Keywords: Morbid Obesity; Laparoscopic Sleeve Gastrectomy; Perioperative Complication; Obesity Surgery Mortality Score; Body Mass Index
MeSH Terms: conditions — Obesity, Morbid | interventions — Reoperation; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Complication positive: Patients with perioeprative complications after laparascopic sleeve gastrectomy before discharge (wound complications, thromboembolic events, staple line leakage, splenic infarction proven by imaging modalities, bleeding detected due to low hemoglobin and hematocrit values during follow-up, acute renal failure due to deterioration in biochemical parameters)
  Interventions: Procedure: Laparascopic Sleeve Gastrectomy; Procedure: İnterventional radiologic drainage; Diagnostic Test: Complte Blood Count and Biochemical evaluation; Diagnostic Test: Computed tomography
- Complication negative: Patients without perioeprative complications after laparascopic sleeve gastrectomy before discharge
  Interventions: Diagnostic Test: Complte Blood Count and Biochemical evaluation
- BMI 40 - 45 kg/m2: Operated patients preoperative BMI values between 40 - 45 kg/m2
  Interventions: Diagnostic Test: Complte Blood Count and Biochemical evaluation
- BMI 45 - 50 kg/m2: Operated patients preoperative BMI values between 45 - 50 kg/m2
  Interventions: Diagnostic Test: Complte Blood Count and Biochemical evaluation
- BMI over 50 kg/m2: Operated patients preoperative BMI values 45 - 50 kg/m2
  Interventions: Diagnostic Test: Complte Blood Count and Biochemical evaluation
- Clavien Dindo Major Complications: 1. Any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic and radiological interventions Acceptable therapeutic regimens are: drugs as antiemetics, antipyretics, analgesics, diuretics and electrolytes and physiotherapy This grade also includes wound infections opened at the bedside
  2. Requiring pharmacological treatment with drugs other than such allowed for grade I complications. Blood transfusions, antibiotics and total parenteral nutrition are also included
  Interventions: Procedure: Laparascopic Sleeve Gastrectomy; Procedure: İnterventional radiologic drainage; Diagnostic Test: Complte Blood Count and Biochemical evaluation; Diagnostic Test: Computed tomography
- Clavien Dindo Minor Complciations: 3. Requiring surgical, endoscopic or radiological intervention 3a Intervention under regional/local anaesthesia 3b Intervention under general anaesthesia 4. Life-threatening complication requiring intensive care/intensive care unit management 4a Single-organ dysfunction 4b Multi-organ dysfunction 5. Patient demise
  Interventions: Procedure: İnterventional radiologic drainage; Diagnostic Test: Complte Blood Count and Biochemical evaluation; Diagnostic Test: Computed tomography

INTERVENTIONS:
Procedure: Laparascopic Sleeve Gastrectomy — Operations performed for complciation of laparascopic sleeve gastrectomy
  Other Names: Reoperation
  Groups: Clavien Dindo Major Complications; Complication positive
Procedure: İnterventional radiologic drainage — İnterventional radiologic drainage of gastric leakage
  Groups: Clavien Dindo Major Complications; Clavien Dindo Minor Complciations; Complication positive
Diagnostic Test: Complte Blood Count and Biochemical evaluation — blood samples obtained from patients to determine the hgb and htc levels of patients and biochemical changes of patients after surgery
Diagnostic Test: Computed tomography — Admitted to observe leakage
  Groups: Clavien Dindo Major Complications; Clavien Dindo Minor Complciations; Complication positive

SUMMARY:
The term obesity is defined as body mass index (BMI) 30 and over, and morbid obesity is considered as BMI greater than 40 (1).Its incidence in the general population is approximately 20% according to Organisation for data of Economic Co-operation and Development (OECD) countries and unfortunately, it is increasing worldwide (2). Obesity should not be thought ofas a single disorderasit is related tomany disorders like hypertension, diabetes, obstructive sleep apnea, cardiovascular diseases, and increased risk of malignancies (1).For years people have struggled with obesitywithboth metabolic and physical problems. Surgical treatment is the most effective long-term therapeutic treatment in current and modern medicine of obesity and obesity-related diseases as the last resort.(3-5). Roux-en-y gastrojejunostomy is the method that has been applied for many years and there isconsensus on its effect.However, in recent years, laparoscopic sleeve gastrectomy (LSG) has an increasing number of procedures with a short learning curve and it is the most performed surgical technique all over the world and also in Turkey (2,6).

Unfortunately, like any surgical procedure, this surgery has its own complications.Although being performed frequently increases the experience of surgeons, this situation cannot reduce the risk of complications of surgery to zero. In morbid obesity patients, the risk of any complications in all surgical procedures is higher than withother patients who were not morbidly obese. Due to these complications, prolonged hospital stays, increased reapplications to the hospital, reoperations and deaths can result(5,7). Despite both an increased risk of complications according to obesity and the risk of specific complications due to sleeve gastrectomy, laparoscopic sleeve gastrectomy is associated with acceptable postoperative morbidity and mortality rates (8).

Various classifications have been described in the literature for complications after surgery.In one of these classifications, according to Clavien-Dindo (CD) Classification, complications are divided into two groups as major and minor. (1, 9)(Table 1). This classification can be applied to bariatric and metabolic surgeries as withall surgery types. Especially major complications in this classification are life-threatening situations and their early detection is important (8).

In fact, surgeons do not want to encounter mortality in any of their patients. In this respect, DeMaria et al. developed an easily applicable mortality risk scoring system, which is consisted of five items (age ≥45 years, male sex, body mass index (BMI) ≥ 50 kg / m2, arterial hypertension, and risk factors for pulmonary thromboembolism) and can be used for the pre-operative determination of risky patients in obesity surgery(Obesity Surgery Mortality Risk Score; OR-MRS) (8,10,11).

In this study, it is aimed to determine the perioperative complications seen in the laparoscopic sleeve gastrectomy patients that we performed in our clinic without being discharged from the hospital and to evaluate the treatment processes of the complications under literature. In addition, whether the OS-MRS risk assessment scale and BMI had a role indetermining perioperative complications before discharge was investigated.

DETAILED DESCRIPTION:
Material - Method Our study was carried out with the approval numbered 13281952-929 from Elazig Training and Research Hospital. All procedures performed in studies involving human participants were in accordance with the ethical standards of the institutional and/or national research committee and with the 1964 Helsinki declaration and its later amendments or comparable ethical standards. 1752 patients who met the criteria of patient selection in terms of obesity and metabolic disease surgery, operated in the Elazığ Training and Research Hospital General Surgery Clinic between January 2016 and October 2018 were evaluated retrospectively. Patients' data were obtained from epicrisis forms in the hospital computer system, patient follow-up charts and patient files. Data for OS-MRS and Clavien Dindo complication classification were obtained from patient follow-up charts, patient files and hospital computer records. Patients' demographic data (age, sex), presence of comorbidities, complications (wound complications, thromboembolic events, leakage from anastomosis, splenic infarction proven by imaging methods, bleeding detected due to low hemoglobin and hematocite values during follow-up, acute renal failure due to deterioration in biochemical parameters) seen in follow up period before discharge (postoperative first 72 hours), complication type (major and minor), whether emergency surgery was performed, BMI values, postoperative hospitalization and OS-MRS. Additionally, while grouping according to BMI values, patients with BMI values below 40 were excluded and three groups with BMI values of 40 - 45 kg / m^2, 45 - 50 kg / m^2 and 50 kg / m^2 and above were created. It was investigated whether there were any complications among these groups and the presence of major or minor complications by CD classification. 1617 patients who met the inclusion criteria were evaluated.

IBM Statistical Package for Social Sciences (SPSS) 20.0 was used for statistical evaluation. Kolmogorow-Smirnov test results were examined in terms of the suitability of the groups for normal distribution. In comparisons between groups, independent sample t-test or Mann Whitney U test was used to evaluate numerical data according to normality test. In the evaluation of categorical data, chi-square analysis and Fischer's exact test were performed. In terms of the relation between complication formation and BMI, univariate analysis and multivariate analysis were performed. Numerical data were given as mean ± standard deviation (ss) (minimum - maximum values) or median (minimum - maximum values) according to normality test. Categorical data are given as count (n) and percentage (%).

ELIGIBILITY:
Inclusion Criteria:

* Patients whose data was available
* Morbid obesity patients who were operated with surgical technique laparoscopic sleeve gastrectomy

Exclusion Criteria:

* Patients whose data was not available
* Patients who were operated with other types of bariatric metabolic surgery
* Patients who left the hospital due to referral
* Patients whose OS-MRS scale wasn't calculated
* Patients whose American Society of Anesthesiologists (ASA) score was 4 or greater

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient selection in terms of obesity and metabolic disease surgery(12);
  1. Patients with a body mass index (BMI) of 40 and above, without the additional comorbid disease,
  2. Patients with a BMI of 35 and above, withtheadditional comorbid disease (such as hypertension, diabetes mellitus)
Sampling Method: Probability Sample
Enrollment: 1617 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Relation between preoperative BMI levels and perioperative complication positivity before discharge | postoperative 72 hour period before discharge
  Relation between preoperative BMI levels and perioperative complication positivity before discharge
Relation between preoperative OS-MRS and perioperative complication positivity before discharge | postoperative 72 hour period before discharge
  Relation between preoperative OS-MRS and perioperative complication positivity before discharge

SECONDARY OUTCOMES:
Perioperative complication rates after laparascopic sleeve gastrectomy before discharge | postoperative 72 hour period before discharge
  Perioperative complication rates after laparascopic sleeve gastrectomy before discharge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Falk V, Twells L, Gregory D, Murphy R, Smith C, Boone D, Pace D. Laparoscopic sleeve gastrectomy at a new bariatric surgery centre in Canada: 30-day complication rates using the Clavien-Dindo classification. Can J Surg. 2016 Apr;59(2):93-7. doi: 10.1503/cjs.016815. PMID 27007089
- [Background] Kirkil C, Aygen E, Korkmaz MF, Bozan MB. QUALITY OF LIFE AFTER LAPAROSCOPIC SLEEVE GASTRECTOMY USING BAROS SYSTEM. Arq Bras Cir Dig. 2018 Aug 16;31(3):e1385. doi: 10.1590/0102-672020180001e1385. PMID 30133677
- [Background] Angrisani L, Santonicola A, Iovino P, Formisano G, Buchwald H, Scopinaro N. Bariatric Surgery Worldwide 2013. Obes Surg. 2015 Oct;25(10):1822-32. doi: 10.1007/s11695-015-1657-z. PMID 25835983
- [Background] van Mil SR, Duinhouwer LE, Mannaerts GHH, Biter LU, Dunkelgrun M, Apers JA. The Standardized Postoperative Checklist for Bariatric Surgery; a Tool for Safe Early Discharge? Obes Surg. 2017 Dec;27(12):3102-3109. doi: 10.1007/s11695-017-2746-y. PMID 28620895
- [Background] Welbourn R, Hollyman M, Kinsman R, Dixon J, Liem R, Ottosson J, Ramos A, Vage V, Al-Sabah S, Brown W, Cohen R, Walton P, Himpens J. Bariatric Surgery Worldwide: Baseline Demographic Description and One-Year Outcomes from the Fourth IFSO Global Registry Report 2018. Obes Surg. 2019 Mar;29(3):782-795. doi: 10.1007/s11695-018-3593-1. Epub 2018 Nov 12. PMID 30421326
- [Background] Chang SH, Freeman NLB, Lee JA, Stoll CRT, Calhoun AJ, Eagon JC, Colditz GA. Early major complications after bariatric surgery in the USA, 2003-2014: a systematic review and meta-analysis. Obes Rev. 2018 Apr;19(4):529-537. doi: 10.1111/obr.12647. Epub 2017 Dec 20. PMID 29266740
- [Background] Major P, Wysocki M, Pedziwiatr M, Malczak P, Pisarska M, Migaczewski M, Winiarski M, Budzynski A. Can the Obesity Surgery Mortality Risk Score predict postoperative complications other than mortality? Wideochir Inne Tech Maloinwazyjne. 2016;11(4):247-252. doi: 10.5114/wiitm.2016.64448. Epub 2016 Dec 6. PMID 28194244
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] DeMaria EJ, Portenier D, Wolfe L. Obesity surgery mortality risk score: proposal for a clinically useful score to predict mortality risk in patients undergoing gastric bypass. Surg Obes Relat Dis. 2007 Mar-Apr;3(2):134-40. doi: 10.1016/j.soard.2007.01.005. PMID 17386394
- [Background] Garcia-Garcia ML, Martin-Lorenzo JG, Liron-Ruiz R, Torralba-Martinez JA, Garcia-Lopez JA, Aguayo-Albasini JL. Failure of the Obesity Surgery Mortality Risk Score (OS-MRS) to Predict Postoperative Complications After Bariatric Surgery. A Single-Center Series and Systematic Review. Obes Surg. 2017 Jun;27(6):1423-1429. doi: 10.1007/s11695-016-2506-4. PMID 27975153
- [Background] Fried M, Yumuk V, Oppert JM, Scopinaro N, Torres A, Weiner R, Yashkov Y, Fruhbeck G; International Federation for Surgery of Obesity and Metabolic Disorders-European Chapter (IFSO-EC); European Association for the Study of Obesity (EASO); European Association for the Study of Obesity Obesity Management Task Force (EASO OMTF). Interdisciplinary European guidelines on metabolic and bariatric surgery. Obes Surg. 2014 Jan;24(1):42-55. doi: 10.1007/s11695-013-1079-8. PMID 24081459